CLINICAL TRIAL: NCT06094205
Title: Understanding and Restoring Speech Production Using an Intracortical Brain-computer Interface
Brief Title: Feasibility of the BrainGate2 Neural Interface System in Persons With Tetraplegia (BG-Speech-02)
Acronym: BG-Speech-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh R. Hochberg, MD, PhD. (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Leigh R. Hochberg, MD, PhD., Neurologist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009p000505 (BG-Speech-02); 1DP2DC021055 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-10-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Anarthria; Dysarthria; Tetraplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Locked-in Syndrome; Muscular Dystrophies
MeSH Terms: conditions — Dysarthria; Quadriplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Locked-In Syndrome; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BrainGate Neural Interface System (Experimental): Placement of the BrainGate2 sensor(s) into the speech-related cortex
  Interventions: Device: BrainGate Neural Interface System

INTERVENTIONS:
Device: BrainGate Neural Interface System — Placement of the BrainGate2 sensor(s) into the speech-related cortex

SUMMARY:
The goal of this study is to improve our understanding of speech production, and to translate this into medical devices called intracortical brain-computer interfaces (iBCIs) that will enable people who have lost the ability to speak fluently to communicate via a computer just by trying to speak.

DETAILED DESCRIPTION:
The goal is to develop a new way to help people who lose the ability to speak due to neurological conditions including ALS or stroke, using an implanted medical device called a "brain-computer interface". The implanted medical device measures the person's brain activity as they try to talk and outputs their intended speech. By bypassing the injured parts of the nervous system this way, we can observe how individual brain cells are involved in speaking and working together as a network, to produce speech, and we can learn to decipher this activity to output what the person is trying to say.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age
* Clinical diagnosis of spinal cord injury, brainstem stroke, muscular dystrophy, amyotrophic lateral sclerosis or other motor neuron disorders
* Complete or incomplete tetraplegia (quadriplegia)
* Must live within a three-hour drive of the Study site and geographically stable for at least 15 months after enrollment.

(There are additional inclusion criteria)

Exclusion Criteria:

* Visual impairment such that extended viewing of a computer monitor would be difficult even with ordinary corrective lenses
* Chronic oral or intravenous steroids or immunosuppressive therapy
* Other serious disease or disorder that could seriously affect ability to participate in the study

(There are additional exclusion criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensor implant duration for at least one-year without any device-related Serious Adverse Events or explant | 1 year
  To determine the safety of the Sensor and overall safety of the System. Participants will be considered a success for this safety measure if they are successfully implanted with the Sensor(s) and:
  1. the sensors are not explanted for safety reasons during the one-year post-implant evaluation period.
  2. there are no device-related Serious Adverse Events that result in death or permanently increased disability during the one-year post-implant evaluation period.

SECONDARY OUTCOMES:
Decoded speech output accuracy | At participant exit from study, or up to 5 years
  The purpose of this feasibility measure is to define the metrics by which a larger trial of intracortical recording for the restoration of speech-based communication might be planned. The secondary endpoints are:
  * The word error rate of speech that is output by the System
  * The phoneme error rate of speech that is output by the System

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Stavisky, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States